CLINICAL TRIAL: NCT01837914
Title: Maxillary Expansion Treatment of Pediatric Obstructive Sleep Apnea
Brief Title: Maxillary Expansion Treatment of Pediatric OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Benjamin Pliska, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H12-02721
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxillary expansion as First treatment (Experimental): Orthodontic expansion of upper jaw, then cross-over to adenotonsillectomy
  Interventions: Procedure: Maxillary expansion; Procedure: Adenotonsillectomy
- Adenotonsillectomy as First treatment (Active Comparator): surgical removal of tonsils and adenoids, then cross-over to maxillary expansion
  Interventions: Procedure: Maxillary expansion; Procedure: Adenotonsillectomy

INTERVENTIONS:
Procedure: Maxillary expansion
Procedure: Adenotonsillectomy

SUMMARY:
Obstructive Sleep Apnea is a serious medical condition affecting an estimated 1-5% of children. The disease is believed to have several overlapping causes including large tonsils and small or narrow jaws. This prospective, randomized cross-over study will evaluate the effectiveness of orthodontic treatment of narrow upper teeth and jaws compared to the current standard of care which is surgical removal of the adenoids and tonsils.

Patients will be evaluated by both an orthodontist and ENT physician, complete a series of questionnaires and undergo an overnight sleep study, both initially and after undergoing the randomized treatment. Patients who on reassessment have residual symptoms of sleep apnea will then be crossed over and receive the other form of treatment. The levels of improvement to both subjective (questionnaire) and objective (overnight sleep study) measures of sleep apnea will then be compared.

The null hypothesis is there is no significant difference in improvement between maxillary expansion and adenotonsillectomy in the objective and subjective outcome measures in children with mild to moderate obstructive sleep apnea.

DETAILED DESCRIPTION:
Background Literature Review Obstructive sleep apnea syndrome (OSAS) is a sleep disorder characterized by recurrent, partial or complete episodes of upper airway obstruction, commonly associated with intermittent hypoxemia and sleep fragmentation.1 The best data available from international studies reports a prevalence rate of 1.2-5.7% in children.2-4 The potential consequences of OSAS in children are serious and include failure to thrive5, attention deficit and hyperactivity disorder6, excessive daytime sleepiness7, and poor learning6. There is also significant concern about long-term cardio-pulmonary risks in these patients8. Not surprisingly, along with higher morbidity, children with OSAS also have higher use of health care services starting from the first year of life9.

OSAS is a multifactorial disease, with the primary cause in children thought to be hypertrophic tonsils and adenoids. However the persistence of OSAS following surgery to remove the tonsils and adenoids is not uncommon. Recent studies using a moderate cut-off apnoea-hyponea index (AHI) of greater than 5 events per hour in relatively low-risk populations, have demonstrated that 13%10 to 29%11 of children have residual OSAS following adenotonsillectomy (AT). Craniofacial form also clearly plays a role in pediatric OSAS as skeletal discrepancies such as transverse maxillary deficiency have been strongly associated with the disease12,13, and skeletal malocclusion has been found to be predictive of a higher AT failure rate14. While the precise nature of the contribution of craniofacial proportions to OSAS remains to be characterized, there is early evidence in the literature to support maxillary expansion (ME) as an alternative treatment to surgery. Results of OSAS treatment with ME have suggested that it may be effective in reducing sleep respiratory disturbances in patients with15 and without16 tonsillar hypertrophy. However, limitations existing in the study designs have left unanswered questions as to the role of ME in the treatment of children suffering from OSAS. Furthermore the studies have been limited to patient populations in Rome, Italy, and while anatomical factors are key determinants of the predisposition to airway collapse, their relative importance for OSAS risk likely varies between ethnicities.17 For this reason, further studies examining these effects on a diverse multicultural population such as that found in North America and in particular urban centers such as Vancouver, Canada are warranted to realize the potential of this novel form of OSAS treatment.

Study Purpose The purpose of this study is to explore the efficacy of maxillary expansion in the treatment of OSAS in children with tonsil and adenoid hypertrophy.

3. Hypothesis The null hypothesis is there is no significant difference in improvement between maxillary expansion and adenotonsillectomy in the objective and subjective outcome measures in children with mild to moderate obstructive sleep apnea.

4. Objectives 4.1: Aim 1- To validate the methodology. The methodology will be validated through conducting this pilot study and analyzing the preliminary data that are generated - if required, improvements in methodology design can be identified during this pilot study to assist in design modification before a larger multi-site study.

4.2: Aim 2- To obtain preliminary data to provide the basis for a larger scale multi-centre randomized controlled trial The results of this study will be analyzed, and if it is under-powered to avoid type II error as predicted from the sample size calculations, the data will used to leverage further funding for a multi-site study.

5. Methods and Statistics 5.1: Research Design Pilot, randomized, controlled single-blinded crossover study. (see Figure 1 - Study Design).

5.2: Study Patient Selection The study patients will be recruited from the Pediatric Otolaryngology Outpatients Clinic and the Pediatric Sleep Disorders Clinic at BC Children's Hospital, with fully informed consent from parents/caregivers and assent from study patients.

Inclusion criteria:

* Ages 5.0 to 10.0 years at the time of screening;
* Diagnosed with obstructive sleep apnea defined as AHI>2, confirmed on overnight, laboratory-based PSG;
* Parental report of witnessed apneas or habitual snoring (on average more than 3 nights per week);
* Deemed to be a candidate for ME by orthodontic evaluation;
* Deemed to be a candidate for tonsillectomy and adenoidectomy by otolaryngologic evaluation.

Exclusion criteria:

* Severe OSA or significant hypoxemia in the presence of tonsillar or adenoid hypertrophy requiring surgical intervention defined as AHI>25 or SpO2 <90% for >2% sleep time.
* An associated craniofacial syndrome or anomaly, including cleft lip and/or palate, or any anatomic or systemic condition that would otherwise exclude the patient from orthodontic treatment.
* Recurrent tonsillitis that meets American Academy of Otolaryngology - Head and Neck Surgery clinical practice guidelines for surgery.
* Extremely overweight defined as a body mass index z-score > 2.99 for age group and sex.
* Severe health problems that could be exacerbated by delayed treatment for OSA, including: severe cardiopulmonary disorders (e.g., cystic fibrosis, congenital heart disease); sickle cell disease; poorly controlled asthma (with > 1 hospitalization in last year); epilepsy requiring medication; diabetes (type 1 or type 2) requiring medication; doctor-diagnosed heart disease or cor pulmonale; or a history of stage II hypertension (HTN) defined as > 99% percentile and/or requiring medication.
* Psychiatric or behavioral disorders that would otherwise exclude the patient from receiving orthodontic treatment

5.3: Intervention Before initiating the intervention the child will undergo overnight polysomnography (PSG), clinical examination by a Pediatric Otolaryngologist and an Orthodontist, as well as a series of validated parental questionnaires relating to sleep habits and quality of life of their child. The intervention period is 4 months with equal numbers of patients being randomized to treatment with either ME or AT.

At the end of the 4-month intervention period all children will be recalled to the Pediatric Obstructive Sleep Apnea Clinic at BC Children's Hospital. Again patients will be examined by the PI Pediatric Otolaryngologist and Orthodontist and undergo a repeat series of examinations, sleep studies and questionnaires in the same fashion as their initial appointment. Patients who present with residual OSAS, defined as an AHI>2, on their follow-up sleep study will be crossed over to the other treatment arm of the study. Treatment protocols will be identical to those described and used in the first phase of the study.

Patients requiring the second intervention will be recalled for a follow-up assessment, repeating the series of data collected at their initial appointment. This will again include overnight polysomnography (PSG), clinical examination by a Pediatric Otolaryngologist and an Orthodontist, as well the parental questionnaires relating to sleep habits and quality of life of their child. (see Figure 1 - Study Design)

Children who still have an abnormal AHI after the second intervention (treatment failures) will be referred to the Sleep Clinic at BC Children's Hospital for further assessment and reviewed by the Pediatric Respirologist for consideration of other levels of obstruction that may require either further surgical intervention or prescribed continuous positive airway pressure (CPAP).

5.4: Primary and Secondary Outcomes

Primary outcome:

Primary outcome measure will be change in AHI between initial and post-intervention overnight PSG. All children will undergo an attended overnight polysomnography (sleep study) at B.C. Children's Hospital Pediatric Sleep Laboratory. The data recorded will include the typical montage monitoring of electroencephalography (EEG), electrooculography (EOG), chin and leg electromyography (EMG), and one electrocardiography (ECG) lead. Respiration is monitored with nasal cannula, mouth thermistor or thermo-couple, thoracic and abdominal bands, finger pulse oxymetry, and neck microphone. Scoring of sleep stages and of respiratory events will follow previously-accepted published guidelines.

The American Academy of Sleep Medicine, the American Academy of Pediatrics, and the American Academy of Otolaryngology all define obstructive sleep apnea as an AHI >1, as calculated by overnight polysomnography. The articles cited in our rationale use a moderate cutoff point of AHI>5 out of convenience in order to highlight their outcome data.

The use of an AHI>2 for the present study is based on a large body of literature, including a recently published outline of an ongoing multi-centered clinical trial (Redline et al. Sleep 2011;34(11):1509) examining the outcomes of surgical treatment of OSA, which also used an AHI>2 as inclusion criteria for the study. A cutoff of 2 is used as a conservative measure to ensure ample justification for treatment. Furthermore, as maxillary expansion treatment is considered less invasive than the standard surgical AT intervention, the inclusion of patients with mild OSAS who might most benefit from non-surgical treatment is justified.

Secondary outcome:

Secondary outcome measures include changes in the Children's Sleep Habits Questionnaire18 (CSHQ), and the OSAS Quality of Life Survey19 (OSA-18) between the initial and post-intervention (4 months) timepoints. The CSHQ is a retrospective 45-item parent reported sleep-screening instrument to delineate sleep habits and identify problematic sleep domains in school-aged children. The CSHQ includes items relating to a number of key sleep domains that encompass the major presenting clinical sleep complaints in this pediatric age group: bedtime behavior and sleep onset; sleep duration; anxiety around sleep; behavior occurring during sleep and night wakings; sleep-disordered breathing; parasomnias; and morning waking/daytime sleepiness. Parents are asked to recall sleep behaviors occurring over a "typical" recent week.39 The OSA-18 is an 18-item questionnaire that uses a Likert-type scoring system to collect information about 5 subscales that are considered to be elements in quality of life: sleep disturbance, physical symptoms, emotional symptoms, daytime function, and caregiver concerns.40 This is also completed by the parent. The Glasgow Children's Benefit Inventory: a new instrument for assessing health-related benefit after an intervention. Ann Otol Rhinol Laryngol. 2004;113(12):980-6). This is a validated instrument specifically designed to measure caregiver satisfaction with a procedural intervention and is ideal for our purpose. This is completed by the parent.

5.5: Randomization The parent or guardian will receive verbal and written detail of the study, and be given the opportunity to consider this information before providing informed consent to participate. If a decision to participate is made, the child will be allocated a study reference number by the study coordinator. Randomization will be based on a pre-established randomization table. To ensure an even distribution of study patient numbers between the groups, patients will be randomized in blocks with blocks sizes randomized between 2 and 4 to prevent identification bias. It is also pre-established that if a child (or their caregiver) decides to opt-out of the study after randomization but before beginning any treatment, the next identified child would be a replacement for the drop-out child with same treatment schedule. If a child dropped out once the any treatment is initiated, there would be no replacement and the subject would be included in the analysis on an intention-to-treat basis.

For children randomized to ME, treatment will begin either at the private dental office of the Principal Investigator or in the Dental Department of BC Children's Hospital. Expansion treatment will be performed by the PI Orthodontist. Additional treatment or referral for comorbidities and education regarding general sleep hygiene and healthy behaviors, and use of nasal saline spray as needed for nasal mucosal crusting or dryness will also be initiated. Costs for orthodontic treatment are not typically covered by the provincial heath insurance plan and therefore will be paid through the operating costs of the study. The ME protocol will follow the standard of care for orthodontic treatment of maxillary constriction. Pre and post-treatment records including lateral and posterior-anterior cephalometric and panoramic radiographs, dental study casts, and intra and extra-oral photos will be collected. An expansion appliance will be bonded to the molar teeth of the upper arch, with a rate of expansion set at 0.25mm each day. A minimum of 7mm of total expansion will be performed. An expansion appliance may be also attached to the lower arch at the discretion of the treating orthodontist should it be indicated by the clinical conditions of the patient. ME patients will have follow up appointments to access the progress of expansion at 2 week intervals for the first month, then monthly until appliance removal 4 months later. Upon removal of the expansion appliance, patients will be provided with a removable dental retainer and then recalled 6 months later for observation as for non-study patients undergoing this form of orthodontic treatment.

For those patients randomized to AT, the procedure will follow the standard of care for this procedure. The AT will be performed by the co-investigator Pediatric Otolaryngologist at the BC Children's Hospital. A standardized technique for tonsillectomy (using bipolar extracapsular dissection) and adenoidectomy (using monopolar suction cautery) will be used. Patients will have the standard peri-operative care, post-operative monitoring, and post-operative follow-up as for non-study patients undergoing this procedure for this indication. Additional treatment or referral for comorbidities and education regarding general sleep hygiene and healthy behaviors, and use of nasal saline spray as needed for nasal mucosal crusting or dryness will also be initiated.

5.6: Blinding Assessment and scoring of the primary (overnight sleep studies) outcome variable will be performed by Dr. David Wensley, director of the BCCH Sleep Lab. Dr. Wensley will be blinded to the treatment received by each patient.

5.7: Sample Size For this pilot study we anticipate recruiting 30 patients, with 15 entering into each initial treatment arm of the study. An informal audit of the referral pattern to the Pediatric Otolaryngology Clinic at BC Children's Hospital has revealed that approximately 15-25 potentially eligible subjects are seen per month. Therefore assuming a very conservative recruitment rate of 5 subjects per month, investigators estimate it may take approximately 6 months to complete subject enrollment,

Drop-out/non-compliance rate:

We estimate a low drop-out rate from the study, based on other studies of this age-group and pathology, and we expect drop-outs to be unrelated to treatment effectiveness, therefore would be randomly distributed between the groups. Assuming a drop-out rate of around 30%, we will require recruitment of 39 study patients to have complete data on 30 study patients.

Study Patient compliance:

To reinforce general study participation, after two months a research assistant will contact via telephone all patients' families to provide advice as well as for safety and adverse event monitoring. At the end of the 4-month intervention period all children will be recalled to BCCH for follow-up examinations and testing.

However due to the invasive nature and inconvenience for children and their family to attend an overnight sleep study at a hospital, recruitment into the study and the possibly required three PSGs may become an issue. To overcome this concern, a patient incentive of $50 per sleep study, to compensate the family for their time and inconvenience as been budgeted.

5.8: Data

Data handling and record keeping:

A study coordinator will be responsible for data collection and storage of randomization codes. The numeric data will be stored electronically using REDCap. All electronic files will be password protected. Information about study patients and study materials will be kept in a locked file cabinet in the Ear, Nose and Throat Clinic at BCCH. The study records will continue to be stored in these lockers 5 years after the study has completed.

Data analysis:

A two-sample t-test will be used to compare groups after randomization into the two treatment arms. Repeated measures ANOVA will be used to evaluate overall treatment effect between initial and follow up data for the primary and secondary outcome measures.

A logistic regression model will be used to relate AHI to combined dental and craniofacial variables. Pearson correlation will measure initial intermolar width, mandibular plane angle and tonsillar score to changes in the PSG parameters, OSA-18 and CSHQ score before and after treatment. Receiver operating characteristic (ROC) curves will be constructed to determine the sensitivity and specificity associated with any given cutoff of the dentofacial variables in predicting PSG diagnosed OSA. For all statistical analyses P < .05 will be considered statistically significant. The results of this pilot study will be underpowered to provide any statistically significant conclusions, however the initial data will be invaluable in future grant applications necessary for larger scale clinical trials, as well as for streamlining patient flow and participation within the Pediatric Obstructive Sleep Apnea Clinic at BCCH. Analysis of this preliminary data will also guide future work to focus on specific measures and outcomes of potential significance.

6. Risk

This study carries no significant safety risk to the participants, beyond the recognized risks of the two interventions:

ME: Minor risks include those associated with undergoing routine and well-established orthodontic treatment for maxillary constriction. As with any intra-oral procedure, there is a risk of aspirating or ingesting materials or instruments, as well as irritation of the soft and hard tissues of the oral cavity. These risks are well understood and generally accepted by patients and parents in the routine delivery of any form of dental or orthodontic care.

AT: Adenoidectomy and tonsillectomy can be associated with post-operative infection or post-operative hemorrhage, sometimes requiring antibiotic administration (<10%), readmission to hospital (<2%), and/or a return to the operating room for hemostatic control (<2%). These risks have low incidence, and are inherent to the surgical procedure, but are not specific to this research study. As adenotonsillectomy is the current standard of care for these subjects, no additional risk is being undertaken to participate in this study if this intervention is included.

The risk of undergoing ME as the first intervention, subsequently failing to improve, and therefore being subject to a minimum 4 month delay before receiving of the current standard of care intervention (AT) - is recognized to have minimal clinical significance in this population of children with non-severe OSA.

7. After the study Study patients will be followed by the Pediatric Otolaryngology Clinic at BC Children's Hospital on an as needed basis, but as a minimum patients will be recalled at 6 months following their completion of the study, or normalization of their symptoms, to assess the long-term improvement to their sleep disordered breathing. This appointment will consist of a clinical exam and general questions to both the patient and parents, as would be standard for any post-treatment follow-up appointment in the Otolaryngology department

8. Difficulties and Limitations The main weakness of the study stems from the fact that it is a pilot project for the interdisciplinary management of children with OSA. Patient flow through the study will require careful monitoring and coordination between three different departments within BCCH.

To maximize efficiency and convenience for participating patients, the PI, Co-Investigator, and study coordinator will meet at least twice monthly to review any adverse events in patient flow through the study or timely delivery of study interventions.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6.0 to 10.0 years at the time of screening;
* Diagnosed with obstructive sleep apnea defined as AHI>2, confirmed on overnight, laboratory-based PSG;
* Parental report of witnessed apneas or habitual snoring (on average more than 3 nights per week);
* Deemed to be a candidate for ME by orthodontic evaluation;
* Deemed to be a candidate for tonsillectomy and adenoidectomy by otolaryngologic evaluation.

Exclusion Criteria:

* Severe OSA or significant hypoxemia in the presence of tonsillar or adenoid hypertrophy requiring surgical intervention defined as AHI>25 or SpO2 <90% for >2% sleep time.
* An associated craniofacial syndrome or anomaly, including cleft lip and/or palate, or any anatomic or systemic condition that would otherwise exclude the patient from orthodontic treatment.
* Recurrent tonsillitis that meets American Academy of Otolaryngology - Head and Neck Surgery clinical practice guidelines for surgery.
* Extremely overweight defined as a body mass index z-score > 2.99 for age group and sex.
* Severe health problems that could be exacerbated by delayed treatment for OSA, including: severe cardiopulmonary disorders (e.g., cystic fibrosis, congenital heart disease); sickle cell disease; poorly controlled asthma (with > 1 hospitalization in last year); epilepsy requiring medication; diabetes (type 1 or type 2) requiring medication; doctor-diagnosed heart disease; or a history of stage II hypertension (HTN) defined as > 99% percentile and/or requiring medication.
* Psychiatric or behavioral disorders that would otherwise exclude the patient from receiving orthodontic treatment

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2013-05; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | 4 months after intervention
  Polysomnography sleep test score

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Pliska, DDS, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Otolaryngology Department, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
NA no IPD will be shared